CLINICAL TRIAL: NCT04702854
Title: Evaluation of Ultrasound Biomicroscopy in the Local Staging of Cutaneous Melanoma
Acronym: BMUMM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-AOIP-04
Record Dates: First submitted 2020-12-02; First posted 2021-01-11 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Cutaneous Melanoma
MeSH Terms: conditions — Melanoma | interventions — Microscopy, Acoustic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Measure of cutaneous melanomas by ultrasound biomicroscopy
  Interventions: Diagnostic Test: Ultrasound Biomicroscopy

INTERVENTIONS:
Diagnostic Test: Ultrasound Biomicroscopy — Measure of cutaneous melanomas by ultrasound Biomicroscopy

SUMMARY:
Cutaneous melanomas represent 4 to 11% of cutaneous cancers, but is responsible for 75% of the deaths reported for these pathologies. The incidence rate double every 10 years. Fourteen thousand cases and 1700 deaths were reported in France in 2015.

The local staging of the cancer is represented by the Breslow index, which is measured on histological analysis, corresponding to the maximum depth of the cancer. Breslow index is a good pronostic value, and is used to choose for the best treatment for the patient.

Having access to the Breslow index before the first resection of the tumor would allow dermatologists to make a complete resection with the best treatment, and the analysis of the sentinel lymph node, all during the same surgical time. Currently, patients need 2 surgeries : one before the Breslow index, and a second one after.

The depth of cutaneous melanoma was already evaluated with High-Frequency Ultrasound (HF-US), but gave disappointing results, with Breslow index not being accurately measured.

Only 50% of tumors less than 2mm depth were efficiently measured. Results were even worst for bigger tumors.

Ultrasound biomicroscopy (UBM) is a new approach, depending on the use of ultra high frequency and large-band transducer. Nice's CHU acquired the only ultrasound device capable of applying such ultra high frequency ultrasound (UHF-US) to human tissues. The device is a VEVO MD (Vevo MD, Toronto, Canada) and equip the Ultrasound Department since June 2018.

The images investigators can assess with this device have an axial resolution of 30µm, for a maximum emission frequency of 70MHz, which was not attainable until this day in human care.

Furthermore, when compared to some of the mono-frequency devices investigators experimented before, this device allow investigators to attain a maximum depth of analysis up to 8mm.

In consequence, this device seems to be able to realize an extremely precise analysis of the skin, and of the cutaneous melanomas, for a structural analysis, as well as a precise depth measurement, and should be evaluated in the measurement of the Breslow Index.

The objective of the study is to analyze the interest of ultrasound biomicroscopy in the pre-therapeutic evaluation of the Breslow index of cutaneous melanoma, compared to histological findings.

The study will include 60 patients with cutaneous melanomas, recently diagnosed in the Dermatology Department of the Nice University Hospital (Pr Bahadoran, Pr Passeron, Pr Lacour). Each patient will beneficiate from complete Ultrasound biomicroscopy analysis of the tumor The examination will be made blindly by 2 operator, both with experience in Ultra High frequency Ultrasound examinations (Dr Azulay, Dr Raffaelli).

The maximum depth of the melanoma (Breslow index) will be recorded in µm. After surgical resection, the histologic analysis (Dr Long, Pr Hofman, Clinical and Experimental AnatomoPathologic laboratory, Nice's University Hospital) will measure the gold-standard Breslow Index.

The comparison will analyze the capacity of Ultrasound biomicroscopy for a precise measurement of the Breslow Index, as well as the inter and intra-operator concordance.

If the results of this study are positives and suggest a modification of the therapeutic strategy, a larger multicentric study would be launched in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of cutaneous melanoma
* Age ≥ 18 years
* Social Security affiliation
* Approval of patient and signature of informed consent form

Exclusion Criteria:

* Counter-indication to the surgical resection of the cutaneous melanoma
* Vulnerable patient (Under-supervision patients or deprived of liberty patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Measurement of the Breslow Index with Ultrasound Biomicroscopy | In the 14 days following the inclusion
  The measurement of the thickness of the malignant melanoma will be carried out in Ultrasound Biomicroscopy in two orthogonal planes using the maximum value obtainedThe measurement will be performed pre-operatively with the device (transducer) attached to an articulated arm from the anterior edge of the lesion to the interface between the posterior border of the lesion and the underlying dermis or hypodermis.
  The measurement will be expressed in mm. The histological measurement will be performed according to the usual techniques after fixation of the surgical specimen. It will also be expressed in µm.

SECONDARY OUTCOMES:
Measurement of the thickness of the malignant melanoma with High Frequency Ultrasound (18MHz) and compare it to the result obtained by Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Conventional High Frequency Ultrasound (18MHz) will be performed prior to Ultrasound Biomicroscopy analysis using an 18 MHz probe according to the usual technique used in High Frequency Ultrasound (freehand) and the thickness of the malignant melanoma will be expressed in µm. Standard gold is defined as at the main objective.
Measurement of the thickness of the malignant melanoma with High Frequency Ultrasound and compare it to the result obtained by Ultrasound Biomicroscopy | In the 14 days following the inclusion
  High Frequency Ultrasound (33MHz) will be performed prior to Ultrasound Biomicroscopy analysis using an 33 MHz probe according to the usual technique used in High Frequency Ultrasound (freehand) and the thickness of the malignant melanoma will be expressed in µm. Standard gold is defined as at the main objective.
Global echogenicity of the malignant melanoma in Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Global echogenicity of the malignant melanoma in relation to the dermis: hypoechoic, isoechoic, hyperechoic
Avascular areas of malignant melanoma using power Doppler in Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Presence of Avascular areas of malignant melanoma using power Doppler in Ultrasound Biomicroscopy Data will be compared with the histological data
Measurement of the thickness of the malignant melanoma with Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Measurement of the thickness of malignant melanoma Ultrasound Biomicroscopy by 2 differents investigators to evaluate the intra and inter-observer matching.
Measurement of the radiofrequency signal acquired during the Ultrasound Biomicroscopy examination of malignant melanoma | In the 14 days following the inclusion
  The radiofrequency signal acquired in Ultrasound Biomicroscopy will be analyzed on a platform dedicated to image processing, looking for radio frequency signal specifics of melanoma, compared to adjacent healthy skin.
Structure of the malignant melanoma in Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Homogeneous or heterogeneous structure of the malignant melanoma in Ultrasound Biomicroscopy
Hyperechoic or anechogenic foci of the malignant melanoma in Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Presence of hyperechoic or anechogenic foci in Ultrasound Biomicroscopy
hyperechoic spans of the malignant melanomain Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Presence of hyperechoic spans in Ultrasound Biomicroscopy
Appearance of the contours of the melanoma | In the 14 days following the inclusion
  Appearance of the contours of the melanoma in Ultrasound Biomicroscopy : regular, irregular, or blurred
Type of vascularization of malignant melanoma using power Doppler in Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Type of vascularization of malignant melanoma using power Doppler in Ultrasound Biomicroscopy: homogeneous, heterogeneous Data will be compared with the histological data
Intensity of vascularization relative to the adjacent normal dermis of malignant melanoma using power Doppler in Ultrasound Biomicroscopy | In the 14 days following the inclusion
  Intensity of vascularization relative to the adjacent normal dermis, with Doppler parameters fixed Data will be compared with the histological data

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas AZULAY, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France